CLINICAL TRIAL: NCT07155954
Title: Value of Super-resolution Ultrasound Microvascular Imaging in Distinguishing Benign and Malignant Superficial Lymph Nodes: a Prospective Multi-center Study
Brief Title: Value of Super-resolution Ultrasonography in Differentiating Benign and Malignant Lymph Nodes
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024853
Record Dates: First submitted 2025-04-07; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-02

CONDITIONS: Lymphadenopathy; Lymphnode Metastasis; Lymphoma; Lymphatic Tuberculosis
MeSH Terms: conditions — Lymphadenopathy; Lymphoma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- benign lymph nodes: the lymph nodes are benign disease proved by pathology
  Interventions: Diagnostic Test: SRUS imaging of the lymph nodes before surgery or biopsy
- malignant lymph nodes: lymph nodes are metastatic lymph nodes or lymphoma proved by pathology
  Interventions: Diagnostic Test: SRUS imaging of the lymph nodes before surgery or biopsy

INTERVENTIONS:
Diagnostic Test: SRUS imaging of the lymph nodes before surgery or biopsy — Ultrasound contrast agent (Sonovue/Sonazoid) is administered to the patients through a peripheral vein. When the micro-bubbles enter the lymph nodes, super-resolution ultrasonography imaging will initiate immediately, to capture the trajectory of the micro-bubbles, thus construct a map of the microvascular distribution.

SUMMARY:
Lymph nodes are one of the most important components of the human immune system, and superficial lymph node enlargement lacks specificity.

Ultrasound examination has been widely used in the diagnosis of lymph node lesions and is of great significance in distinguishing between benign and malignant. However, the two-dimensional and Doppler ultrasound features of different types of lymph node lesions overlap and intersect, and the blood flow perfusion information of lymph nodes can provide more information for differentiation.

At present, the widely used contrast-enhanced ultrasound is easier to evaluate blood flow perfusion and can display small blood vessels smaller than 100 microns. The diagnostic accuracy of cervical lymph nodes using contrast-enhanced ultrasound is 80-90%.

However, current contrast-enhanced ultrasound is limited by physical diffraction, with a resolution ranging from sub-millimeter to millimeter. This limitation hinders the visualization of small blood vessels or microcirculation by ultrasound, and parameters such as vascular size, spatial vascular pattern, and velocity of microcirculation are crucial for disease diagnosis and prognosis evaluation. Super resolution ultrasound (SRUS) is a new blood flow imaging technique. By tracking the movement trajectory of micro-bubbles instead of imaging the micro-bubbles themselves, the ultrasound diffraction limit can be exceeded to improve the sensitivity and image resolution of blood flow.

Thus the study aim to evaluate the feasibility of SRUS technology in distinguishing between benign and malignant lymph nodes, and compare the differences in blood flow distribution and perfusion index between benign and malignant lymph nodes under SRUS imaging.

DETAILED DESCRIPTION:
The study aim to evaluate the feasibility of SRUS technology in distinguishing between benign and malignant lymph nodes, and compare the differences in blood flow distribution, perfusion index, CEUS parameters, blood supply mode between benign and malignant lymph nodes under SRUS imaging.

ELIGIBILITY:
Inclusion Criteria:

* (1)suggested abnormal lymph nodes indicated by ultrasonography; (2) Patients scheduled for lymph nodes puncture or fine needle aspiration or surgery; (3) Age greater than or equal to 18 years old.

Exclusion Criteria:

* (1) Pregnant and lactating women; (2)pathological results not indicating benign or malignant lymph nodes; (3) history of chemotherapy or radiotherapy ; (4) History of allergies to eggs, milk, and ultrasound contrast agents; (5) Patients with acute coronary syndrome, severe pulmonary hypertension, or acute respiratory distress syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abnormal lymph nodes and who are scheduled for lymph nodes puncture or fine needle aspiration or surgery
Sampling Method: Non-Probability Sample
Enrollment: 779 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-10-22 (Estimated); Study Completion 2027-10-22 (Estimated)

PRIMARY OUTCOMES:
benign or malignant pathology results from biopsy or surgery | within 1 month after SRUS imaging

SECONDARY OUTCOMES:
The expression level of various immuno-histochemical indicators of lymph nodes | within 2 months after SRUS imaging
Microvascular Quantitative Indices between benign and malignant lymph nodes by SRUS | within 2 months after the SRUS
Microvascular Quantitative Indices between lymph node metastasis and lymphoma | within 2 months after the SRUS imaging
Blood supply mode of CEUS between benign and malignant lymph nodes | within 2 months after the SRUS imaging
Quantitative analysis parameters of CEUS between benign and malignant lymph nodes | within 2 months after SRUS imaging
  Quantitative analysis parameters of CEUS including AT, TTP, PKI, MTT, and AUC between benign and malignant lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: li g cui, Chief Physician, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided